CLINICAL TRIAL: NCT01736917
Title: Phase II Study of Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone in Patients With Germ Cell Tumors Undergoing 5 Day Cisplatin-based Chemotherapy: Hoosier Oncology Group Study QL12-153
Brief Title: Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone in Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lawrence Einhorn (Other)
Collaborators: Hoosier Cancer Research Network (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Lawrence Einhorn, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL12-153
Record Dates: First submitted 2012-11-21; First posted 2012-11-29 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
Keywords: Fosaprepitant; 5HT3 Receptor Antagonists; Dexamethasone; Germ Cell Tumors; Testis Cancer; Rescue Medications
MeSH Terms: conditions — Vomiting; Neoplasms, Germ Cell and Embryonal; Testicular Neoplasms | interventions — fosaprepitant; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone (Experimental): Patients must have no nausea and/or vomiting for 24 hours and must not have used other anti-emetics for 72 hours prior to starting protocol treatment. Treatment must not start until this criteria is satisfied.
  * Any germ cell chemotherapy regimen utilizing Cisplatin (20mg/m2 x 5 days).
  Acute emesis prophylaxis:
  * Any 5HT3 receptor antagonist may be used D1 - 5 or D1, 3 and 5 if palonosetron is used per institutional standards.
  * Dexamethasone 20mg PO (orally) daily, D1 and 2
  * Fosaprepitant 150mg IV on day 3
  Delayed emesis prophylaxis:
  * Fosaprepitant 150mg IV on D5
  * Dexamethasone 4mg PO BID (twice a day) on D6, 7 and 8
  PRN antiemetics allowed at the discretion of the treating investigator
  * No additional doses of 5HT3 receptor antagonist, dexamethasone, or fosaprepitant will be given during the acute or delayed treatment periods
  Interventions: Drug: Fosaprepitant; Drug: Dexamethasone; Drug: 5HT3

INTERVENTIONS:
Drug: Fosaprepitant — Fosaprepitant 150mg IV D3 for acute prophylaxis Fosaprepitant 150mg IV on Day 5 for delayed prophylaxis
Drug: Dexamethasone — Dexamethasone 20mg PO daily on D1 and 2 for acute prophylaxis Dexamethasone 4mg PO BID on Days 6 through 8
Drug: 5HT3 — Any 5HT3RA on D1-5; D1, 3 and 5 if palonosetron is used.

SUMMARY:
The hypothesis is that the substitution of multi-day oral aprepitant with (intravenous) IV fosaprepitant, in combination with a 5-HT3 receptor antagonists (5HT3RA) + dexamethasone will provide comparable protection from 5 day cisplatin chemotherapy induced nausea and vomiting, compared to the results of our prior study of aprepitant. This study will be the first clinical trial evaluating fosaprepitant in patients receiving multi-day cisplatin. This will be a single arm, phase II study. The investigators propose to utilize intravenous (IV) fosaprepitant on days 3 and 5 of the 5-day cisplatin chemotherapy regimen. It is anticipated that fosaprepitant can suppress delayed chemo-induced nausea and vomiting for 2-5 days after therapy. This study will test the value of fosaprepitant in this patient population.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Treatment Regimen:

Patients must have no nausea and/or vomiting for 24 hours and must not have used other anti-emetics for 72 hours prior to starting protocol treatment. Treatment must not start until this criteria is satisfied.

Any germ cell chemotherapy regimen utilizing cisplatin (20mg/m^2 x 5 days). This will usually be combined with bleomycin (BEP), etoposide (EP), ifosfamide (VIP), vinblastine (VeIP), paclitaxel (TIP) or epirubicin. All of these regimens get the identical cisplatin, which is the only highly emetic drug in any of the chemo regimens.

Acute emesis prophylaxis (administered per institutional standards prior to chemotherapy):

* Any 5HT3 receptor antagonist may be used days 1 through 5 or days 1, 3 and 5 if palonosetron is used per institutional standards.
* Dexamethasone 20mg PO (orally) daily, days 1 and 2
* Fosaprepitant 150mg IV on day 3

Delayed emesis prophylaxis:

* Fosaprepitant 150mg IV on day 5
* Dexamethasone 4mg PO BID (twice a day) on days 6, 7 and 8

PRN (as needed) antiemetics allowed at the discretion of the treating investigator

* No additional doses of 5HT3 receptor antagonist, dexamethasone, or fosaprepitant will be given during the acute or delayed treatment periods

ECOG Performance Status of 0-2

Life Expectancy: Not specified

Hematopoietic:

* White blood cell count (WBC) > 3.0 K/mm3
* Absolute neutrophil count ≥ 1.5 K/mm3
* Hemoglobin (Hgb) > 10 g/dL
* Platelets > 100 K/mm3

Hepatic:

* Bilirubin < 1.5 x ULN (upper limit of normal)
* Aspartate aminotransferase (AST, SGOT) ≤ 3 x ULN
* Alanine aminotransferase (ALT, SGPT) ≤ 3 x ULN

Renal:

* Creatinine ≤ 2 mg/dl

ELIGIBILITY:
Inclusion Criteria:

* Male patients ≥15 years of age with histologically or cytologically confirmed diagnosis of germ cell tumor receiving a standard 5 day cisplatin based chemotherapy regimen. Prior chemotherapy is allowed. Patients do not have to be chemo naïve.
* Written informed consent and HIPAA authorization for release of personal health information.
* Patients must have had no nausea or vomiting for 24 hours and no anti-emetic use for 72 hours prior to starting protocol therapy. Treatment must not start in registered patients until this criteria is met.

Exclusion Criteria:

* No active central nervous system (CNS) metastases. Patients with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis. NOTE: A patient with prior brain metastasis may be considered if they have completed their treatment for brain metastasis, no longer require corticosteroids, and are asymptomatic.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, Gleason < grade 7 prostate cancers, or other cancer for which the patient has been disease-free for at least 1 year.
* No previous treatment with any investigational agent within 30 days prior to registration for protocol therapy.
* No concurrent participation in a clinical trial which involves another investigational agent.
* No use of agents expected to induce the metabolism of fosaprepitant which include: rifampin, rifabutin, phenytoin, carbamazepine, and barbiturates.
* No concurrent use of agents which may inhibit metabolism of fosaprepitant which include: cisapride, macrolide antibiotics (erythromycin, clarithromycin, azithromycin), azole antifungal agents (ketoconazole, itraconazole, voriconazole, fluconazole), amifostine, nelfinavir, calcium channel antagonists such as verapamil and diltiazem, and ritonavir.
* No concurrent use of warfarin while on study.
* No known history of anticipatory nausea or vomiting.
* No clinically significant infections as judged by the treating investigator.

Min Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Einhorn, M.D., Study Chair — Hoosier Cancer Research Network
Locations (4):
- United States (4):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Siteman Cancer Center, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - MUSC Hollings Cancer Center, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costantine Albany, Nasser H. Hanna, Joel Picus, Ralph J. Hauke, Christopher A. Fausel, Ziyue Liu, Mary J. Brames, Lawrence H. Einhorn. Phase II study of fosaprepitant plus 5HT3 receptor antagonists plus dexamethasone in patients with germ cell tumors undergoing 5-day cisplatin-based chemotherapy: Hoosier Oncology Group QL12-153. J Clin Oncol 32:5s, 2014 (suppl; abstr TPS4594)
- [Result] Brames MJ, Case-Eads S, Hanna NH, Fausel CA, Breen T, Einhorn LH. Phase II study of fosaprepitant +5HT3 receptor antagonist + dexamethasone in patients with germ cell tumors undergoing 5-day cisplatin-based chemotherapy: A Hoosier Cancer Research Network Study. J Clin Oncol 33:5s, 2015 (suppl; abstr e20737)
- [Derived] Adra N, Albany C, Brames MJ, Case-Eads S, Johnson CS, Liu Z, Fausel CA, Breen T, Hanna NH, Hauke RJ, Picus J, Einhorn LH. Phase II study of fosaprepitant + 5HT3 receptor antagonist + dexamethasone in patients with germ cell tumors undergoing 5-day cisplatin-based chemotherapy: a Hoosier Cancer Research Network study. Support Care Cancer. 2016 Jul;24(7):2837-42. doi: 10.1007/s00520-016-3100-y. Epub 2016 Feb 2. PMID 26838019
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone: Patients must have no nausea and/or vomiting for 24 hours and must not have used other anti-emetics for 72 hours prior to starting protocol treatment. Treatment must not start until this criteria is satisfied.
  - Any germ cell chemotherapy regimen utilizing Cisplatin (20mg/m^2 x 5 days).
  Acute emesis prophylaxis:
  * Any 5HT3 receptor antagonist may be used D1 - 5 or D1, 3 and 5 if palonosetron is used per institutional standards.
  * Dexamethasone 20mg PO (orally) daily, D1 and 2
  * Fosaprepitant 150mg IV on day 3
  Delayed emesis prophylaxis:
  * Fosaprepitant 150mg IV on D5
  * Dexamethasone 4mg PO BID (twice a day) on D6, 7 and 8
  PRN antiemetics allowed at the discretion of the treating investigator
  * No additional doses of 5HT3 receptor antagonist, dexamethasone, or fosaprepitant will be given during the acute or delayed treatment periods
  Fosaprepitant: Fosaprepitant 150mg IV D3 for acute prophylaxis Fosaprepitant 150mg IV on Day 5 for delayed prophyl
Period: Overall Study
Arm/Group | Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone
Started | 65
Completed | 54
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 10

BASELINE CHARACTERISTICS:
Population: 64 participants were consented and treated per protocol. 1 participant listed in participant flow experienced an adverse event during infusion and was immediately taken off study. His baseline characteristics are not included in this table.
Arm/Group | Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 33 [15 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 64
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 64
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  participants
    ECOG PS 0 | 59
    ECOG PS 1 | 4
    ECOG PS 2 | 1
Cancer Stage [Number; unit: participants] — Stage 0 Abnormal cells are present but have not spread to nearby tissue. Also called carcinoma in situ, or CIS. CIS is not cancer, but it may become cancer.
  Stage I, Stage II, and Stage III Cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Stage IV The cancer has spread to distant parts of the body.
  participants
    Cancer Stage I | 27
    Cancer Stage II | 24
    Cancer Stage III | 11
    Cancer Stage IS | 1
    Cancer Stage Unknown | 1
Prior Chemotherapy [Number; unit: participants]
  Participants with Prior Chemotherapy | 5
  Participants without Prior Chemotherapy | 59
Chemotherapy Regimen [Number; unit: participants]
  Bleomycin, etoposide, cisplatin | 51
  Etoposide, cisplatin | 10
  Vinblastine, ifosfamide, cisplatin | 2
  Cisplatin, Epirubicin | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response of Acute and Delayed Chemotherapy Induced Nausea and Vomiting
Description: complete response (CR) of both acute (days 1 through 5) and delayed (days 6 through 8) CINV, defined by no emetic episodes or use of rescue medications
Time Frame: Days 1-8 of chemotherapy regimen
Measure: Number; unit: percentage of participants
Groups:
- Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone: Patients must have no nausea and/or vomiting for 24 hours and must not have used other anti-emetics for 72 hours prior to starting protocol treatment. Treatment must not start until this criteria is satisfied.
  * Any germ cell chemotherapy regimen utilizing Cisplatin (20mg/m2 x 5 days).
  Acute emesis prophylaxis:
  * Any 5HT3 receptor antagonist may be used D1 - 5 or D1, 3 and 5 if palonosetron is used per institutional standards.
  * Dexamethasone 20mg PO (orally) daily, D1 and 2
  * Fosaprepitant 150mg IV on day 3
  Delayed emesis prophylaxis:
  * Fosaprepitant 150mg IV on D5
  * Dexamethasone 4mg PO BID (twice a day) on D6, 7 and 8 PRN antiemetics allowed at the discretion of the treating investigator
  * No additional doses of 5HT3 receptor antagonist, dexamethasone, or fosaprepitant will be given during the acute or delayed treatment periods Fosaprepitant: Fosaprepitant 150mg IV D3 for acute prophylaxis Fosaprepitant 150mg IV on Day 5 for delayed prophyl
Arm/Group | Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone
Number analyzed (Participants) | 54
percentage of participants
  acute phase(days 1 through 5) | 29.6
  delayed phase (days 6 through 8) | 46.3
  overall | 24.1

2. Secondary Outcome: Total Number of Emetic Episodes
Description: total number of emetic episodes
Time Frame: Days 1-8 of chemotherapy regimen
Measure: Number; unit: episodes
Arm/Group | Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone
Number analyzed (Participants) | 54
episodes | 29

3. Secondary Outcome: Use of Rescue Medications.
Description: Total number of patients who received rescue medications.
Time Frame: Days 1-8 of chemotherapy regimen
Measure: Number; unit: participants
Groups:
- Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone: Patients must have no nausea and/or vomiting for 24 hours and must not have used other anti-emetics for 72 hours prior to starting protocol treatment. Treatment must not start until this criteria is satisfied.
  - Any germ cell chemotherapy regimen utilizing Cisplatin (20mg/m2 x 5 days).
  Acute emesis prophylaxis:
  * Any 5HT3 receptor antagonist may be used D1 - 5 or D1, 3 and 5 if palonosetron is used per institutional standards.
  * Dexamethasone 20mg PO (orally) daily, D1 and 2
  * Fosaprepitant 150mg IV on day 3
  Delayed emesis prophylaxis:
  * Fosaprepitant 150mg IV on D5
  * Dexamethasone 4mg PO BID (twice a day) on D6, 7 and 8
  PRN antiemetics allowed at the discretion of the treating investigator
  * No additional doses of 5HT3 receptor antagonist, dexamethasone, or fosaprepitant will be given during the acute or delayed treatment periods
  Fosaprepitant: Fosaprepitant 150mg IV D3 for acute prophylaxis Fosaprepitant 150mg IV on Day 5 for delayed prophyl
Arm/Group | Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone
Number analyzed (Participants) | 54
participants | 37

4. Secondary Outcome: Self-Reported Assessment of Nausea
Description: the patient's self-reported assessment of nausea Days 1-8 using a 0-100mm visual analog scale (VAS) median.
  The Visual Analouge (VAS) 100mm Scale Score for Chemotherapy Induced Nausea and Vomiting (CINV). Participants were asked to mark a linear scale 100mm in length representing their level of nausea with 0mm indicating no nausea and 100mm indicating severe nausea. Median VAS scores (in mm) are reported, per day.
Time Frame: Days 1-8 of chemotherapy regimen
Population: 54 patients completed the VAS on all 8 days and were eligible for analysis.
Measure: Median (Full Range); unit: millimeters
Arm/Group | Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone
Number analyzed (Participants) | 54
millimeters
  median VAS score - day 1 | 0 [0 to 24]
  median VAS score - day 2 | 0 [0 to 76]
  median VAS score - day 3 | 4.5 [0 to 60]
  median VAS score - day 4 | 18.5 [0 to 95]
  median VAS score - day 5 | 23.5 [0 to 92]
  median VAS score - day 6 | 12.5 [0 to 80]
  median VAS score - day 7 | 7 [0 to 90]
  median VAS score - day 8 | 3 [0 to 84]

ADVERSE EVENTS:
Time Frame: Duration of participation on study, up to 8 days.
Arm/Group | Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 9/65
Other Adverse Events (participants affected / at risk) | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone (N=65)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosaprepitant + 5HT3 Receptor Antagonists + Dexamethasone (N=65)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (7)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (4)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (2)
ALLERGIC REACTION (Immune system disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 14 (14)
ANEMIA (Blood and lymphatic system disorders) | 13 (21)
ANOREXIA (Metabolism and nutrition disorders) | 19 (26)
ANXIETY (Psychiatric disorders) | 9 (11)
AORTIC VALVE DISEASE (Cardiac disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2)
AZOOSPERMIA (Reproductive system and breast disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (6)
BLOATING (Gastrointestinal disorders) | 4 (4)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
CHILLS (General disorders) | 3 (4)
CHOLESTEROL HIGH (Investigations) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 17 (19)
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 (11)
CREATININE INCREASED (Investigations) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 8 (10)
DIZZINESS (Nervous system disorders) | 5 (6)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 24 (29)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 9 (9)
EDEMA LIMBS (General disorders) | 4 (5)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1)
FATIGUE (General disorders) | 53 (78)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FEVER (General disorders) | 7 (7)
FLUSHING (Vascular disorders) | 5 (5)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 11 (11)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 10 (15)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 14 (15)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOT FLASHES (Vascular disorders) | 2 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 5 (10)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (2)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 4 (9)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (7)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPONATREMIA (Metabolism and nutrition disorders) | 5 (10)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 3 (4)
INR INCREASED (Investigations) | 1 (5)
INSOMNIA (Psychiatric disorders) | 13 (13)
LOCALIZED EDEMA (General disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 5 (9)
MALAISE (General disorders) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 10 (11)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 53 (90)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
NEUTROPHIL COUNT DECREASED (Investigations) | 14 (27)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2)
ORAL PAIN (Gastrointestinal disorders) | 2 (2)
PAIN (General disorders) | 14 (14)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
PARESTHESIA (Nervous system disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 4 (4)
PLATELET COUNT DECREASED (Investigations) | 8 (14)
PRESYNCOPE (Nervous system disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 5 (5)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 6 (6)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SINUS PAIN (Nervous system disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 2 (3)
SOMNOLENCE (Nervous system disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 4 (5)
SYNCOPE (Nervous system disorders) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 8 (9)
TOOTHACHE (Gastrointestinal disorders) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (2)
URINARY FREQUENCY (Renal and urinary disorders) | 2 (2)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 9 (9)
WEIGHT GAIN (Investigations) | 8 (8)
WHITE BLOOD CELL DECREASED (Investigations) | 13 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No